CLINICAL TRIAL: NCT07101887
Title: Comparative Study Between the Use of Trapeziometacarpal Prostheses and the Usual Resection-tenosuspension Arthroplasty for the Treatment of Rhizarthrosis.
Brief Title: Comparative Study Between the Use of Trapeziometacarpal Prostheses and the Usual Resection-tenosuspension Arthroplasty for the Treatment of Rhizarthrosis, Focusing on Changes in Pain (Measured With the VAS Scale) and Function (With the Quick-DASH).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/8942/I
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-02

CONDITIONS: Rizarthrosis
Keywords: Thumb; osteoarthritis; prosthesis; trapeziectomy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maia Prosthesis group (Experimental)
  Interventions: Procedure: Implantation of thumb prosthesis
- Trapeziectomy and Burton-Pellegrini technique (Experimental): Remove the trapezium bone and perform a suspensionplasty using a hemi-slip of the flexor carpi radialis tendon
  Interventions: Procedure: Burton-Pellegrini technique

INTERVENTIONS:
Procedure: Implantation of thumb prosthesis — Replacing the articular surface of the trapezo-metacarpal joint with a socked-ball prosthesis.
  Arms: Maia Prosthesis group
Procedure: Burton-Pellegrini technique — Remove the trapezium bone and perform a suspensionplasty using a hemi-slip of the flexor carpi radialis tendon
  Arms: Trapeziectomy and Burton-Pellegrini technique

SUMMARY:
It is a randomized, prospective, single-blind study of two treatment techniques for rhizarthrosis. The patients are divided into two groups: one in which a Maia trapeziometacarpal prosthesis is implanted, and the other in which the standard technique of trapeziectomy and tenosuspension plasty is performed according to the Burton-Pellegrini technique.The follow-up of the patients is one year, and functionality (measured with the Quick Dash test) and pain (measured with the VAS scale) are compared throughout this period.This study has a sample size of 62 patients, 31 per group. Other secondary variables are also evaluated, such as strength and mobility of the thumb trapeziometacarpal joint (measured with the Kapandji index).

ELIGIBILITY:
Inclusion Criteria:

* Rizarthrosis grade I, II, III

Exclusion Criteria:

* Rizarthrosis grade IV
* Severe osteoporosis
* Metals allergy
* Previous surgical interventions related
* Malformations in the articular zones that difficult the implant placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
VAS | 1 year
  Pain evaluated by Visual analogic scale (VAS)
Quick Dash | 1 year
  Function of the arm evaluated by Quick Dash scale

SECONDARY OUTCOMES:
Strength | 1 year
  Strength evaluated with a pressure gauge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No